CLINICAL TRIAL: NCT01745510
Title: Efficacy of Enteral Administration of the Docosahexaenoic Acid on Necrotizing Enterocolitis, Cytokines and Hospital Stay in Preterm Neonates
Brief Title: Enteral Administration of Docosahexaenoic Acid to Prevent Necrotizing Enterocolitis in Preterm Neonates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Mariela Bernabe García, Principal investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DHA-ECN; DHA, ECN and Preterm (Other Grant/Funding Number: CONACYT 161643)
Record Dates: First submitted 2012-11-23; First posted 2012-12-10 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Necrotizing Enterocolitis
Keywords: docosahexaenoic acid; n-3 fatty acids; necrotizing enterocolitis; preterm infants
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: The intervention was the docosahexaenoic acid, a nutraceutical derived from the omega 3 fatty acids.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Intervention was blinded through assinging a code, printed and saved into opaque envelopes did it by a researcher who did not participate in the fieldwork.
  Randomization was carried out through the Random Allocation Software v.1
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA Group (Experimental): DHA Group will receive 75 milligrams of docosahexaenoic acid (DHA) per kilogram of their baseline weight.
  They will receive one dose, administered by enteral feeding every 24 h during 14 days
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- Control Group (Placebo) (Placebo Comparator): Control group will receive sunflower oil which is the excipient of the DHA in this study.
  They will receive one dose every 24 h during 14 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — Docosahexaenoic acid from algae source
  Other Names: n-3 Fatty Acids
  Arms: DHA Group
Dietary Supplement: Placebo — Placebo was designed to mimic the color and consistence of the oil that contains DHA
  Other Names: Sunflower oil, Placebo for DHA intervention
  Arms: Control Group (Placebo)

SUMMARY:
* The purpose of this study is to determine whether docosahexaenoic acid is effective in the prevention or reducing severity of necrotizing enterocolitis (NEC) in preterm neonates < 1500 g at birth who are starting enteral feeding.
* if NEC is prevented, this study will measure whether hospital stay is also reduced in neonates who receive Docosahexaenoic acid (DHA)

DETAILED DESCRIPTION:
* Preterm neonates with birth weight less than 1500 g are in higher risk to develop NEC.
* NEC is an inflammatory condition that:

  1. Is the medical urgency most frequent of gastrointestinal tube that requires neonatal intensive care
  2. may perforate infant´s bowel requiring surgery from 20% to 60% of the cases
  3. may cause infant's death in 20% to 42% of the cases.
  4. has no adequate treatment worldwide, therefore prevention is needed
* DHA by enteral feeding has been administrated by our research group to attenuate inflammatory response in septic and surgical neonates.
* Our results showed:

  1. lower Interleukin(IL)-1 beta in septic neonates, but in surgical neonates, they also showed less IL-6 and anti-inflammatory cytokines IL-10 and IL-1ra, after adjusting by confounders
  2. increased weight, length and fat mass gain in septic neonates
  3. decreased organic failures in surgical neonates, and
  4. lower stay at neonatal intensive care in surgical neonates

DHA has not been used as unique intervention at a high but physiological dose; in addition, our previous results found an anti-inflammatory effect in neonates.Therefore, we expect that preterm infants may have a reduced bowel inflammatory response and lower NEC events and or severity

ELIGIBILITY:
Inclusion Criteria:

* Birth weight lower than 1500 g
* Adequate weight for gestational age
* Clinically stable to begin enteral feeding
* Written informed consent by both parents plus the sign of two witnesses

Exclusion Criteria:

* Clinical and biochemical data of inflammatory response such as body core temperature altered, cardiac and respiratory frequency -low or high according to age-, leucocytosis or leucopenia, taking into account the thresholds reported by Goldstein in Pediatric Critical Care Medicine 2005 Vol 6 N°1.
* Persistent bleeding at any level
* Mother taking n-3 supplements and planning to breastfed
* Parents who decline the authorization for participating in the study
* Early discharge to other hospital outside the metropolitan area
* Persistent vomiting
* Receiving medication to avoid coagulation
* Gastrointestinal malformations

Ages: 60 Minutes to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2012-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Necrotizing enterocolitis (NEC) | Patients will be followed for the duration of hospital stay, an expected average of 6 weeks
  Neonates will receive enteral DHA at beginning of their first enteral feeding and NEC will be diagnosed during hospital stay, measured as presence or absence, as well as severity of NEC by Bell's score.

SECONDARY OUTCOMES:
Cytokines Interleukin (IL)-1 beta, Tumoral necrosis factor (TNF)-alpha, IL-6, IL-10 | At baseline and a second measurement only if they develop confirmed or severe NEC according to Bell's criteria
  Plasma cytokines will be determined before to the beginning of the enteral feeding (baseline) and if the infant develop confirmed or severe NEC. Cytokines will be measured by a multiplex kit in picograms/mL.
Hospital stay | The duration of hospital stay, an expected average of 6 weeks
  Hospital stay includes intensive stay care and preterm service (where clinically stable babies are attended) until they are discharged from the hospital to home, in days.
Growth velocity in weight | Throughout hospital stay as part of nutritional follow-up of the care unit, an expected average of 4 weeks
  Gain of weight in g/kd/day, measured with an electronic scale every week until hospital discharge or 40 weeks of corrected gestational age
Growth velocity in length and head circumference | Throughout hospital stay as part of nutritional follow-up of the care unit, an expected average of 4 weeks
  Gain of recumbent length and and head circumference in cm/week measured every 2 weeks until hospital discharge or 40 weeks of corrected gestational age. For measuring length we will use an infantometer and for head circumference we will use a glass fiber tape.
Growth velocity in skin folds | Throughout hospital stay as part of nutritional follow-up of the care unit, an expected average of 4 weeks
  Gain of bicipital, tricipital, suprailiac and subscapular skin folds in mm/week measured every 2 weeks, until hospital discharge or 40 weeks of corrected gestational age. We will use a glass fiber tape to measure it.
Enteral tolerance | During their hospital stay until reach 150 ml/kg/day, in average 2 to 5 weeks
  Registration of volume of the enteral intake every 24 h (ml/kg/day) until reach 150 ml/kg/day and being sustained or increased by enteral feeding with human milk or formula.
Enteral intolerance | During their hospital stay until reach 150 ml/kg/day, in average 2 to 5 weeks
  Registration of number of patients with clinical signs of intolerance such as vomit, abnormal number of stool loss, abdominal distension, number of patients with medical indication to withdraw enteral feeding due clinical unstability and number of patients with use of medications related to enteral tolerance such as omeprazole, ranitidine, vitamins, iron, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Bernabe-Garcia, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Unit of Medical Research in Nutrition, Pediatric Hospital, IMSS, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
This project has secondary outcomes that have not been analyzed; therefore, in this moment we decided not to share our database.

REFERENCES:
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, Del Prado M, Rivera D, Ruiz G, Maldonado J, Villegas R. Docosahexaenoic acid administered in the acute phase protects the nutritional status of septic neonates. Nutrition. 2006 Jul-Aug;22(7-8):731-7. doi: 10.1016/j.nut.2006.04.002. Epub 2006 Jun 5. PMID 16750345
- [Background] Lopez-Alarcon M, Bernabe-Garcia M, del Valle O, Gonzalez-Moreno G, Martinez-Basilea A, Villegas R. Oral administration of docosahexaenoic acid attenuates interleukin-1beta response and clinical course of septic neonates. Nutrition. 2012 Apr;28(4):384-90. doi: 10.1016/j.nut.2011.07.016. Epub 2011 Nov 12. PMID 22079797
- [Background] Bernabe-Garcia M, Lopez-Alarcon M, Villegas-Silva R, Mancilla-Ramirez J, Rodriguez-Cruz M, Maldonado-Hernandez J, Chavez-Rueda KA, Blanco-Favela F, Espinoza-Garcia L, Lagunes-Salazar S. Beneficial Effects of Enteral Docosahexaenoic Acid on the Markers of Inflammation and Clinical Outcomes of Neonates Undergoing Cardiovascular Surgery: An Intervention Study. Ann Nutr Metab. 2016;69(1):15-23. doi: 10.1159/000447498. Epub 2016 Jul 9. PMID 27394149
- [Result] Bernabe-Garcia M, Calder PC, Villegas-Silva R, Rodriguez-Cruz M, Chavez-Sanchez L, Cruz-Reynoso L, Mateos-Sanchez L, Lara-Flores G, Aguilera-Joaquin AR, Sanchez-Garcia L. Efficacy of Docosahexaenoic Acid for the Prevention of Necrotizing Enterocolitis in Preterm Infants: A Randomized Clinical Trial. Nutrients. 2021 Feb 17;13(2):648. doi: 10.3390/nu13020648. PMID 33671220